CLINICAL TRIAL: NCT06653998
Title: Feasibility and Safety of Early Mobilization and Rehabilitation in Intensive Care Unit Patients. A Prospective, Multicenter Study
Brief Title: Feasibility and Safety of Early Mobilization and Rehabilitation in Intensive Care Unit Patients
Status: Recruiting | Type: Observational
Sponsor: Claudia Aristizábal (Other)
Responsible Party: Sponsor-Investigator, Claudia Aristizábal, Director, Sanitas University
Organization: Sanitas University (Other)
Other Study IDs: Motionlife Study
Record Dates: First submitted 2024-10-08; First posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Intensive Care Unit Acquired Weakness; Intensive Care Unit Patients
Keywords: Intensive Care Units; Muscle Weakness; Early Mobilization; Rehabilitation
MeSH Terms: conditions — Muscle Weakness | interventions — Early Ambulation; Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intensive care unit patients: Patients aged ≥ 18 years admitted to intensive care units and receiving the institutional early mobilisation protocol.
  Interventions: Other: Early mobilization and rehabilitation

INTERVENTIONS:
Other: Early mobilization and rehabilitation — In the initial assessment will be applied the ICU Mobility Scale, with the objective of establishing the patient's current level of function and determining the most appropriate type, intensity and duration of activity.
  The sessions, which will be conducted by a physiotherapist, will include therapeutic strategies such as bed exercises (both active and passive), electrical stimulation, use of an in-bed cycloergometer (for upper and lower limbs), sitting on the edge of the bed, bed transfers, bedside transfers from bed to chair, out-of-bed exercises, standing, and walking. The latter two activities are considered to be the most complex. Each session will last approximately 20 to 30 minutes and will be conducted once a day, on a daily basis throughout the patient's ICU stay. The last session wil be prior to discharge of the patient.
  During each session, the Borg Perception of Exertion Scale will be assessed in order to adjust the intensity of physical activity.

SUMMARY:
Intensive Care Unit Acquired Weakness (ICU-AW) is a common complication of critical illnesses, occurring in approximately 50% of ICU patients and is strongly associated with increased morbidity, physical impairments, and both short- and long-term mortality. The main characteristics of ICU-AW are symmetrical generalised muscle weakness affecting both respiratory and limb muscles; however, the clinical phenotype may differ depending on age, disease burden, length of ICU stay, and mechanical ventilation duration.

The objective of the present study is to evaluate the feasibility achieved and the safety outcomes reported in a cohort of critically ill patients who undergo early mobilisation and rehabilitation in intensive care units. This research is a multicentre prospective cohort study.

DETAILED DESCRIPTION:
Prolonged immobilisation, mechanical ventilation, and sedation during critical illness have been associated with generalized muscle weakness, restricted joint mobility, pressure ulcers, critical illness neuropathies or acquired weakness, deep vein thrombosis (DVT), prolonged mechanical ventilation, psychological disorders, and cognitive impairment. Barriers to early mobilisation have been identified, including patient-related, institution-related, and physician-related barriers, and various strategies have been used to overcome these barriers and facilitate the smooth practice of early mobilisation.

Early mobilisation, initiated within 24-48 hours of Intensive Care Unit (ICU) admission, has been shown to be the best strategy for reducing ICU-acquired weakness (ICUAW). It includes a variety of interventions: passive for non-cooperative patients (e.g., positioning, passive joint mobilisation) and active-assisted or active for less or fully cooperative patients (e.g., active or active-assisted joint mobilisation, sitting on bed or chair, transfers, standing, ambulation). Several studies have provided evidence that progressive early mobilisation of adult ICU patients is feasible, safe, and can yield benefits including improved functional outcomes and reduced ICU and hospital stay durations.

Successful implementation of an early physical rehabilitation program in most ICUs requires a structured process to promote quality improvement. This involves a multidisciplinary approach including hospital administrators, ICU and rehabilitation leaders who support the program and promote a culture change within the ICU. It also requires assembling a multidisciplinary team including intensivists, nursing, clinical nutrition, physical medicine, and rehabilitation; establishing a common goal and shared expectation of early rehabilitation for all patients with focused efforts to identify and overcome barriers to achieving this goal; and obtaining basic equipment to facilitate early rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age admitted to the intensive care units.

Exclusion Criteria:

* Patients requiring extracorporeal membrane oxygenation (ECMO).
* Patients without indication for early mobilisation in the ICU (severe hemodynamic instability, acute brain or spinal injury with rest orders, anaemia (Hb <8 mg/dl), thrombocytopenia (platelets <50,000), active systemic inflammatory response according to institutional protocols).
* Patients in the postoperative period of cardiac transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ≥ 18 years of age admitted to the intensive care units of Clínica Reina Sofía, Clínica Universitaria Colombia, Clínica Reina Sofia and Clínica Santa María del Lago in Bogotá.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2024-05-10 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Viability | During the intervention period commenced on the first day of admission to the ICU through study completion, an average of seven days.
  This is the number of sessions performed by the patient.
Safety event | During the intervention period commenced on the first day of admission to the ICU through study completion, an average of seven days.
  This is the number of safety events related with the intervention. The following safety events will be measured: Accidental removal of central venous catheter, accidental removal of endotracheal tube, accidental removal of arterial line, accidental removal of nasogastric or orogastric tube, accidental removal of bladder catheter, high or low blood pressure, tachycardia, bradycardia, arrhythmia, y polypnoea.

SECONDARY OUTCOMES:
Degree of ability achieved | During the intervention period commenced on the first day of admission to the ICU through study completion, an average of seven days.
  It will be assessed using the ICU Mobility Scale.

OTHER OUTCOMES:
Heart rate | During the intervention period commenced on the first day of admission to the ICU through study completion, an average of seven days.
  It will be measured with pulse oximeter.
Respiratory rate | During the intervention period commenced on the first day of admission to the ICU through study completion, an average of seven days.
  It will be measured with pulse oximeter.

CONTACTS AND LOCATIONS:
Locations (4):
- Colombia (4):
  - Clínica Reina Sofia Pediátrica y Mujer, Bogotá, Bogota D.C.
  - Clinica Univesitaria Colombia, Bogotá, Bogota D.C.
  - Clínica Infantil Santa María del Lago, Bogotá, Bogota D.C.
  - Clínica Reina Sofia, Bogotá, Bogota D.C.

REFERENCES:
- [Derived] Parada-Gereda HM, Merchan-Chaverra R, Medina-Parra J, Benavides-Cruz J, Gaitan-Duarte H. Safety of early mobilisation in the intensive care unit: a prospective and multicentre cohort study protocol. BMJ Open. 2025 Aug 26;15(8):e101772. doi: 10.1136/bmjopen-2025-101772. PMID 40858383